CLINICAL TRIAL: NCT07135401
Title: Optimizing MRI Liver Imaging: Evaluating Breath-Holding Techniques and Oxygen Supplementation to Reduce Respiratory Motion Artifacts
Brief Title: Optimizing Liver MRI Using Breath-Holding With and Without Oxygen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 25-44459
Record Dates: First submitted 2025-08-06; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: MRI; MRI Image Enhancement
Keywords: abdominal MRI; breath-hold technique; functional residual capacity; image quality; non-contrast MRI; liver MRI; end-expiration; preoxygenation; oxygen supplementation; radiology; respiratory motion control; T2-weighted imaging; living liver donor; motion artifact; 3T MRI; UCSF; motion artifact reduction; hyperventilation; end-inspiration
MeSH Terms: conditions — Hyperventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Residual Capacity/End-Expiration Without Oxygen (Experimental): Participants will undergo abdominal MRI scans while performing breath-holding at end-expiration without oxygen supplementation. T2-weighted and MRCP sequences will be acquired during breath-hold trials.
  Interventions: Diagnostic Test: Breath-hold conditions
- Functional Residual Capacity/End-Expiration With Oxygen (Experimental): Participants will undergo abdominal MRI scans while performing breath-holding at end-expiration with oxygen supplementation administered prior to. T2-weighted and MRCP sequences will be acquired during breath-hold trials.
  Interventions: Diagnostic Test: Breath-hold conditions

INTERVENTIONS:
Diagnostic Test: Breath-hold conditions — Functional Residual Capacity/End-Expiration (breath-hold technique) with/without oxygen to optimize MRI image quality.

SUMMARY:
The goal of this interventional study (clinical trial) is to learn if different breath-holding techniques, with and without extra oxygen, can improve the quality of abdominal Magnetic Resonance Imaging (MRI) images in healthy adults, ages 18-75.

The main questions it aims to answer are:

* Does breath-holding at end-expiration improve image quality in abdominal MRI scans?
* Does adding oxygen while breath-holding further reduce motion artifacts in abdominal MRI scans?

Researchers will compare breath-holding with and without oxygen to see if using oxygen improves image quality during MRI scans.

Participants will:

* Be pre-screened for MRI safety and trained on breath-hold procedures
* Have one non-contrast abdominal MRI scan at the University of California San Francisco (UCSF) China Basin Imaging Center
* Use two different breath-holding techniques during the scan, with and without oxygen
* Complete one study visit lasting about 45 minutes to 1 hour

DETAILED DESCRIPTION:
This is a within-subject, randomized crossover interventional study conducted at UCSF China Basin Imaging Center using a 3 Tesla Magnetic Resonance Imaging (3T MRI scanner). The study aims to optimize abdominal MRI protocols by evaluating the impact of breath-holding techniques, with and without oxygen supplementation, on motion artifacts and overall image quality.

Each participant will undergo non-contrast abdominal MRI scans using two breath-hold conditions: (1) Functional Residual Capacity (FRC)/end-expiration without oxygen and (2) FRC/end-expiration with preoxygenation. The order of these conditions will be randomized to control for potential order effects, and each participant will serve as their own control to reduce inter-individual variability.

T2-weighted and Magnetic Resonance Cholangiopancreatography (MRCP) sequences will be acquired during each breath-hold trial. MRI-compatible pulse oximetry will be used to monitor oxygen saturation and pulse rate throughout scanning. A radiology research nurse will be present if additional monitoring is needed based on the participant's pre-screening or intra-scan findings. Participants will receive training on breath-hold procedures prior to imaging to improve consistency and comfort during scanning.

Two board-certified radiologists, blinded to the breath-hold condition, will independently assess each image set for motion artifacts and overall image quality using a standardized 5-point grading system. The grading will range from very poor (1) to very good (5) based on sharpness, visibility of anatomical details, and presence of blurring or signal loss.

Inter-rater reliability will be evaluated using the Intraclass Correlation Coefficient (ICC). Statistical analyses will include repeated measures ANOVA to compare image quality scores across breath-holding conditions. Descriptive analyses will assess breath-hold durations and participant characteristics (e.g., age, gender) in relation to image quality and safety outcomes, including oxygen saturation and self-reported comfort.

This study involves minimal risk, does not utilize contrast agents, and is intended to support the development of motion-reduced, efficient liver MRI protocols, particularly for living liver donor evaluation. Data collected during the study will not be used for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be within 18-75 years of age;
* Subject must be able to hear and understand instructions without assistive devices;
* Subject must provide written informed consent;
* Subject has the necessary mental capacity to understand instructions, and is able to comply with protocol requirements;
* Subject is able to remain still for duration of imaging procedure (approximately 30-45 minutes)

Exclusion Criteria:

* Subjects with a weight greater than 499 lbs;
* Subjects that have metallic/conductive or electrically/magnetically active implants without Magnetic Resonance (MR) Safe or Magnetic Resonance (MR) Conditional labeling, with the exception of dental devices/fillings, surgical clips, and surgical staples determined to be safe for MRI scanning by a physician investigator;
* Subjects that have implants with MR Unsafe labeling;
* Subjects that have implants labeled as MR Conditional by the manufacturer for which the allowable conditions are not expected to be achieved by the MR environment or scan protocol;
* Subjects who have a contraindication to MRI per the screening policy of the participating site;
* Subjects with any respiratory or cardiovascular condition that could compromise safe breath holding;
* Subjects who are female and pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Liver MRI Image Quality (Motion Artifacts) | During the single MRI session (approximately 1 hour)
  Image quality of liver MRI scans will be assessed by quantifying the degree of respiratory motion artifacts under two breath-holding conditions: Functional Residual Capacity (FRC) alone and FRC with oxygen supplementation. Reduced artifacts indicate improved image clarity and feasibility of the technique.
  Unit of Measure: Motion artifact score (ordinal scale, e.g., 1-5).

SECONDARY OUTCOMES:
Breath-Holding Duration | During the MRI session (approximately 1 hour)
  The duration (in seconds) that participants can comfortably sustain a breath-hold under each condition (FRC alone and FRC with oxygen supplementation). Unit of Measure: Seconds.
Oxygen Saturation During Breath-Holding | During the MRI session (approximately 1 hour)
  Peripheral oxygen saturation will be monitored during each breath-hold condition to assess physiologic tolerance and safety. Unit of Measure: Percent oxygen saturation (%).
Adverse Events and Participant-Reported Discomfort | During and immediately after the MRI session (up to 1 hour)
  Number and type of adverse events, as well as participant-reported discomfort, occurring during or immediately after each breath-hold condition. Unit of Measure: Number of events.

CONTACTS AND LOCATIONS:
Overall Officials: John P Roberts, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoo JL, Lee CH, Park YS, Kim JW, Lee J, Kim KA, Seol HY, Park CM. The Short Breath-Hold Technique, Controlled Aliasing in Parallel Imaging Results in Higher Acceleration, Can Be the First Step to Overcoming a Degraded Hepatic Arterial Phase in Liver Magnetic Resonance Imaging: A Prospective Randomized Control Study. Invest Radiol. 2016 Jul;51(7):440-6. doi: 10.1097/RLI.0000000000000249. PMID 26807896
- [Background] Vu KN, Haldipur AG, Roh AT, Lindholm P, Loening AM. Comparison of End-Expiration Versus End-Inspiration Breath-Holds With Respect to Respiratory Motion Artifacts on T1-Weighted Abdominal MRI. AJR Am J Roentgenol. 2019 May;212(5):1024-1029. doi: 10.2214/AJR.18.20239. Epub 2019 Mar 5. PMID 30835515
- [Background] Towell V, Gysen KV, Cross S, Kk Low G. Efficacy of preoxygenation administration in volunteers, in extending the end-expiration breath-hold duration for application to abdominal radiotherapy. Tech Innov Patient Support Radiat Oncol. 2023 May 4;26:100208. doi: 10.1016/j.tipsro.2023.100208. eCollection 2023 Jun. PMID 37207259
- [Background] Parkes MJ, Green S, Stevens AM, Parveen S, Stephens R, Clutton-Brock TH. Safely prolonging single breath-holds to >5 min in patients with cancer; feasibility and applications for radiotherapy. Br J Radiol. 2016 Jul;89(1063):20160194. doi: 10.1259/bjr.20160194. PMID 27168468
- [Background] Khot R, McGettigan M, Patrie JT, Feuerlein S. Quantification of gas exchange-related upward motion of the liver during prolonged breathholding-potential reduction of motion artifacts in abdominal MRI. Br J Radiol. 2020 Feb 1;93(1106):20190549. doi: 10.1259/bjr.20190549. Epub 2019 Dec 10. PMID 31778311
- [Background] Funk E, Anderzen-Carlsson A, Ingverud P, Leander A, Thunberg P. Patient-initiated breath-holds in MRI: an alternative for reducing respiratory artifacts and improving image quality. Clin Imaging. 2015 Jul-Aug;39(4):619-22. doi: 10.1016/j.clinimag.2014.12.007. Epub 2014 Dec 13. PMID 25555833
- [Background] Chandarana H, Feng L, Ream J, Wang A, Babb JS, Block KT, Sodickson DK, Otazo R. Respiratory Motion-Resolved Compressed Sensing Reconstruction of Free-Breathing Radial Acquisition for Dynamic Liver Magnetic Resonance Imaging. Invest Radiol. 2015 Nov;50(11):749-56. doi: 10.1097/RLI.0000000000000179. PMID 26146869